CLINICAL TRIAL: NCT07271797
Title: Comparing Different Electronic Apex Locators and Periapical Radiography on Postoperative Pain: A Randomized Clinical Study
Brief Title: Comparing Different Electronic Apex Locators and Periapical Radiography on Postoperative Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20210816
Record Dates: First submitted 2025-11-16; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Acute Pain
Keywords: electronic apex locator; working length; postoperative pain; root canal therapy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Randomized, single-centre endodontic trial; single visit treatment; differeant electronic apex locators.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: In this single-blind clinical trial, participants were unaware of which electronic apex locator was used during root canal treatment. The operator performing the procedure knew the device allocation, but the postoperative pain data were collected by an independent investigator who was blinded to the device used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group 1 (Experimental): Identifies patients who underwent root canal treatment using Root ZX (Morita Corp., Tokyo, Japan)
  Interventions: Device: Root ZX (Morita Corp., Tokyo, Japan)
- Group 2 (Experimental): Identifies patients who underwent root canal treatment using Propex Pixi (Dentsply Maillefer, Ballaigues, Switzerland)
  Interventions: Device: Propex Pixi (Dentsply Maillefer, Ballaigues, Switzerland)
- Group 3 (Experimental): Identifies patients who underwent root canal treatment using Woodpex III (Woodpecker Medical Instrument Co., Guilin, China)
  Interventions: Device: Woodpex III (Woodpecker Medical Instrument Co., Guilin, China)
- Group 4 (Experimental): Identifies patients who underwent root canal treatment using Raypex 6 (VDW, Munich, Germany)
  Interventions: Device: Raypex 6 (VDW, Munich, Germany)
- Group 5 (Experimental): Describe patients who underwent root canal treatment using periapical radiography.
  Interventions: Device: periapical radiography

INTERVENTIONS:
Device: Root ZX (Morita Corp., Tokyo, Japan) — Root ZX (Morita Corp., Tokyo, Japan) is a well-established electronic apex locator widely used in endodontics for determining working length during root canal procedures. It operates based on the ratio method and has been shown to provide reliable and accurate measurements even in the presence of various irrigants. Root ZX has been extensively validated in clinical and laboratory studies and is considered a gold standard among apex locators.
  Arms: Group 1
Device: Propex Pixi (Dentsply Maillefer, Ballaigues, Switzerland) — Propex Pixi (Dentsply Maillefer, Ballaigues, Switzerland) is a compact electronic apex locator designed to determine the working length of root canals with high accuracy. It uses advanced multi-frequency technology to detect the position of the apical foramen and provides real-time feedback through visual and audible signals. Despite its small size, Propex Pixi has demonstrated reliable performance in various clinical settings.
  Arms: Group 2
Device: Woodpex III (Woodpecker Medical Instrument Co., Guilin, China) — Woodpex III (Woodpecker Medical Instrument Co., Guilin, China) is an electronic apex locator that operates using dual-frequency impedance technology to determine the working length of root canals. It features a user-friendly interface with visual and audible indicators, making it suitable for routine clinical use. While it is considered a cost-effective alternative to premium apex locators, studies have shown variable accuracy depending on canal conditions and the presence of irrigants.
  Arms: Group 3
Device: Raypex 6 (VDW, Munich, Germany) — Raypex 6 (VDW, Munich, Germany) is a modern electronic apex locator that utilizes multi-frequency technology to accurately detect the apical constriction during root canal procedures. It features a color-coded graphical display and audible signals to guide clinicians throughout the procedure. Raypex 6 has been reported to provide reliable working length measurements even under challenging clinical conditions.
  Arms: Group 4
Device: periapical radiography — Working length determination using periapical radiography involves placing a small endodontic file inside the root canal and taking a radiograph to estimate the position of the file tip relative to the root apex. This traditional technique is widely used but may be limited by image distortion, anatomical variations, and the two-dimensional nature of radiographs. Despite its limitations, it remains a common reference method in endodontic practice.
  Arms: Group 5

SUMMARY:
This clinical study was conducted to better understand whether the method used to measure the length of root canals affects the amount of pain patients feel after root canal treatment. Accurate measurement of the root canal is important to clean and fill the tooth properly. If the canal is cleaned too short or too far, it may cause discomfort or reduce the success of the treatment.The study included 125 adult patients who had deep decay but no current pain or swelling. All had single-rooted teeth diagnosed with asymptomatic irreversible pulpitis. Participants were randomly divided into five groups, each using a different method to measure the root canal length before treatment. Four of the methods used electronic devices (called apex locators), and one used a dental X-ray. None of the patients knew which method was used in their case, and all treatments were done by the same dentist in a single appointment.Pain levels were recorded using a simple pain scale called the Visual Analog Scale (VAS), where patients marked their pain level at 6, 12, 24, and 48 hours after treatment. Patients were also allowed to take painkillers if needed, and they were asked to record how many tablets they used.The study also looked at factors like age, gender, the location of the treated tooth, and use of pain medication. The study was carried out at Bezmialem Vakif University's Department of Endodontics. All participants gave written consent, and the study was approved by the university's ethics committee. No complications or serious side effects were reported during or after the treatment.

DETAILED DESCRIPTION:
This clinical study aimed to investigate whether the method used to determine root canal length has an effect on postoperative pain following root canal treatment. Accurate measurement of the root canal is crucial for successful cleaning and sealing of the root system. If the measurement is too short or too long, it may lead to discomfort or compromise treatment outcomes.

The study enrolled 125 adult patients who had deep dental caries but were not experiencing any active pain or swelling at the time of diagnosis. All patients had single-rooted teeth diagnosed with asymptomatic irreversible pulpitis, a condition in which the pulp is irreversibly damaged but does not yet cause symptoms. Eligible participants were randomly assigned to one of five groups, each using a different method for working length determination prior to treatment. Four groups used electronic apex locators (Root ZX, Propex Pixi, Woodpex III, and Raypex 6), while one group used periapical radiography (dental X-ray). Treatments were carried out by the same experienced clinician during a single appointment. Patients were blinded to the method used in their treatment.

To evaluate postoperative discomfort, pain levels were assessed using the Visual Analog Scale (VAS), a 10-centimeter scale where patients mark their pain level ranging from "no pain" to "worst imaginable pain." VAS scores were recorded at 6, 12, 24, and 48 hours after treatment. Patients were allowed to take over-the-counter pain medication (400 mg ibuprofen) if necessary, and they were instructed to record how many tablets they took each day.

In addition to pain levels, the study evaluated other potential contributing factors such as patient age, gender, the location of the treated tooth (upper or lower jaw), and use of analgesics. The data were analyzed to determine whether these factors were associated with differences in pain perception among groups.

This study was conducted at the Department of Endodontics, Faculty of Dentistry, Bezmialem Vakif University (Istanbul, Türkiye). Written informed consent was obtained from all participants, and the study protocol was approved by the university's ethics committee. No adverse events or complications were reported during or after the procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following criteria to be included in the trial:
* Aged between 18 and 60 years.
* Diagnosed with asymptomatic irreversible pulpitis in a single-rooted tooth and scheduled for primary root canal treatment in that tooth.
* In good general health, with no systemic diseases.
* No use of any analgesic medications within the last 24 hours prior to the treatment.
* Willing to participate in the study and able to give informed consent.

Exclusion Criteria:

* Patients who do not meet the above inclusion criteria excluded from the study. In other words, any patient outside the specified age range, with systemic health issues, having taken pain medication recently, or without an asymptomatic single-rooted tooth diagnosis as described, not enrolled. Additionally, patients who decline to participate or who cannot provide informed consent excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 125 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Postoperative pain intensity | 6, 12, 24, 48 hours after root canal treatment
  Patient-reported pain intensity on the 10-cm Visual Analog Scale (VAS), where 0 represents "no pain" and 10 represents "worst imaginable pain." Higher scores indicate greater pain intensity. Pain levels were recorded by each participant in a diary. The analysis compares mean VAS scores among groups treated with different electronic apex locators.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakıf University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No